CLINICAL TRIAL: NCT05607524
Title: Effects of Grape King Bio Probiotic Capsules in Promoting Fat Excretion by Human Trial
Brief Title: Effects of Probiotic Capsules in Promoting Fat Excretion by Human Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Principal Investigator, Chin-Lin Hsu, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS2-22068
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Probiotic capsules, 500 mg each, two daily for a total of 1000 mg for 4 weeks
  Interventions: Dietary Supplement: probiotics
- Placebo (Placebo Comparator): The placebo capsules had the same composition as the experimental capsules, except that they did not contain probiotics, and should be used for 4 weeks.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotics — Eat a capsule for once, and twice a day
  Arms: Probiotics
Dietary Supplement: placebo — Eat a capsule for once, and twice a day
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy of 2 capsules (500 mg per capsule, 1000 mg per day) of Grape King Probiotic Capsules per day in promoting fat excretion in obese patients by clinical human food test.

DETAILED DESCRIPTION:
This experiment is carried out in a controlled manner. Before the subjects enter the research experiment, they need to follow their original lifestyle. The habits of maintaining a constant body weight for more than 2 weeks before the test, such as calorie balance in the diet and the amount of activity. Then enter the test to carry out the evaluation test of probiotics to the end. 60 subjects were randomized, 20 to placebo and 40 to probiotics. The subjects took two capsules of Grape King probiotics daily, a total of 1000 mg. Continue to take it for 4 weeks, and perform blood routine tests. Body composition detection, waist and hip circumference measurement, related index analysis and 24-hour dietary questionnaires, gut health questionnaires and stool samples were collected and analyzed for 4 weeks before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* male or female participants
* aged 20-40 years old
* body mass index in 25-27 kg/m2
* body fat > 25% for men and > 30% for women

Exclusion Criteria:

* cancer, chronic heart disease, use drugs which pharmacological effects may affect immunity
* having systemic infections
* using probiotics.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2022-12-29 (Estimated); Study Completion 2023-01-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline fecel lipid weight at week 4 | Week0, Week4
  Compared the difference of fecel lipid weight level between the week 4 and 0

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jou Chien, PhD student, Principal Investigator — Chung Shan Medical University; Xin-Bei Lin, MS student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan